CLINICAL TRIAL: NCT00825266
Title: The Effect of Bosentan and Pioglitazone on Insulin Resistance in Pulmonary Arterial Hypertension
Brief Title: Insulin Resistance in Pulmonary Arterial Hypertension
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: difficulty in finding eligible subjects
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Roham T. Zamanian, Principle Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SU-09052008-1295; IRB#7432
Record Dates: First submitted 2009-01-16; First posted 2009-01-21 (Estimated); Results first posted 2017-03-31 (Actual); Last update posted 2017-03-31 (Actual); Status verified 2017-02

CONDITIONS: Hypertension, Pulmonary
Keywords: pulmonary hypertension & insulin resistance
MeSH Terms: conditions — Hypertension, Pulmonary; Insulin Resistance | interventions — Bosentan; Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- bosentan (Active Comparator): Bosentan 62.5 twice daily for 4 weeks, then 125 mg twice daily.
  Interventions: Drug: bosentan
- Pioglitazone (Active Comparator): Pioglitazone 15 mg a day for 4 weeks then Pioglitazone 30 mg a day for the duration of the study.
  Interventions: Drug: Pioglitazone

INTERVENTIONS:
Drug: bosentan — Bosentan 62.5 mg BID for 4 weeks, then 125mg BID for duration of study.
  Other Names: Tracleer
  Arms: bosentan
Drug: Pioglitazone — Pioglitazone 15 mg a day for 4 weeks then Pioglitazone 30 mg a day for the duration fo the study.
  Other Names: Actos
  Arms: Pioglitazone

SUMMARY:
The purpose of this study is to evaluate 1) the incidence of insulin resistance (a pre-diabetic state) in patients with pulmonary hypertension, and 2) test the utility of a validated PH therapy (Tracleer) versus Pioglitazone in the treatment of those patients found to have insulin resistance.

DETAILED DESCRIPTION:
The Effect of Bosentan and Pioglitazone on Insulin Resistance in Pulmonary Arterial Hypertension ,is a study evaluating the incidence of insulin resistance in patients with pulmonary hypertension and testing the utility of a validated PH therapy(Tracleer) versus Pioglitazone in the treatment of those patients found to have insulin resistance.Patients with PAH must be stable on therapy for at least 3 months are considered for enrollment in this study.With the exception of PAH, subjects must be free of major medical illnesses, including diabetes mellitus ,malignancy or significant hepatic or renal disease.

ELIGIBILITY:
Inclusion Criteria:

Patients with Pulmonary Arterial Hypertension (PAH) must be stable on therapy for at least 3 months prior to enrollment in the trial. We will include patients with idiopathic PAH and Familial PAH as well as PAH associated with collagen vascular disease or drug or toxin exposure. With the exception of PAH, subjects must be free of major medical illnesses, including diabetes mellitus (must have fasting plasma glucose < 126 mg/dL and taking no anti-hyperglycemic agent), malignancy or significant hepatic or renal disease. Subjects may be hypertensive and on anti-hypertensive medications as long as blood pressure is < 150/100 mm Hg. Subjects may also be dyslipidemic and/or taking drugs to improve abnormalities of lipid metabolism, but they will be excluded if they are taking medications known to alter insulin sensitivity, including glucocorticoids, niacin, anti-retrovirals, thiazolidinediones, or metformin. Use of oral contraceptives or estrogen and/or progesterone replacement therapy is permitted. Weight must be stable and the subjects agree not to change their eating habits or exercise regimen during the study period. There will be no restrictions with regard to race or socioeconomic status, and the racial/ethnic composition of the study population will be reflective of the communities surrounding the Stanford University Medical Center.

Exclusion Criteria:

* Vulnerable subject status.

* Concurrent Endothelin-1 antagonist therapy
* Concurrent Thiazolidinedione therapy
* New York Heart Class III or IV
* PAH related to other etiologies.
* Diabetes Mellitus with Fasting Glucose Levels > 126 mg/dL
* Allergy or hypersensitivity to pioglitazone or bosentan administration.
* Current treatment with statin therapy.
* Initiation of PAH therapy (prostacyclin analogues, phosphodiesterase-5 inhibitors) within three months of enrollment.
* Inability or unwillingness to avoid systemic steroid containing medications for four months. Inhaled steroid use is acceptable.
* Current or recent use or planned treatment with: glyburide, cyclosporine, nilotinib, nisoldipine, ranolazine, thioridazine
* Hepatic transaminases > 2x the upper limit of normal at the center at screening.
* Current or recent (< 6 months) chronic heavy alcohol consumption.
* Current use of another investigational drug (non-FDA approved) for PAH.
* Lung transplant recipients.
* History of myositis.
* Renal failure (Cr 2.0).
* Hospitalized or acutely ill.
* Chronic liver disease (cirrhosis, chronic hepatitis, etc.).
* Abnormalities of the arm or hand or radical mastectomy (preventing brachial artery ultrasound).
* Pregnant or lactating women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2008-09; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roham T. Zamanian, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Bosentan: Bosentan 62.5 twice daily for 4 weeks, then 125 mg twice daily.
  bosentan: Bosentan 62.5 mg twice daily for 4 weeks, then 125mg BID for duration of study.
- Pioglitazone: Pioglitazone 15 mg a day for 4 weeks then Pioglitazone 30 mg a day for the duration of the study.
  Pioglitigone: Pioglitazone 15 mg a day for 4 weeks then Pioglitazone 30 mg a day for the duration fo the study.
Period: Overall Study
Arm/Group | Bosentan | Pioglitazone
Started | 1 | 1
Completed | 1 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bosentan | Pioglitazone | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Continuous [Mean (Full Range); unit: years] | 61 [61 to 61] | 51 [51 to 51] | 56 [51 to 61]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Insulin Resistance Profile Change - Triglyceride:HDL Cholesterol Ratio
Description: insulin resistance measured -triglyceride: HDL cholesterol ratio measures at 16 weeks compared with baseline.
Time Frame: baseline and 16 weeks
Measure: Number; unit: ratio
Arm/Group | Bosentan | Pioglitazone
Number analyzed (Participants) | 1 | 1
ratio | -0.22 | -1.96

2. Secondary Outcome: 6 Minute Walk Test
Description: 6 minute walk test measures the distance that a patient can walk on a flat, hard surface in a period of 6 minutes.It assess the disease severity of the subject at 16 week compared to the baseline.
Time Frame: Baseline and 16 weeks
Measure: Number; unit: meters
Arm/Group | Bosentan | Pioglitazone
Number analyzed (Participants) | 1 | 1
meters | -71 | -23

3. Secondary Outcome: NYHA (New York Heart Association Classification) Changes
Description: New York Heart Classification(NYHA) changes measured at 16 weeks compared with baseline.
  NYHA Classification:
  NYHA class I:no symptoms and no limitation in ordinary physical activity NYHA class II:Mild symptoms (mild shortness of breath and/or angina) and slight limitation during ordinary activity NYHA class III:Marked limitation in activity due to symptoms, even during less-than-ordinary activity, NYHA class IV:Severe limitations. Experiences symptoms even while at rest. {Higher NYHA class represent worse symptoms}
Time Frame: Baseline and 16 weeks
Measure: Number; unit: NYHA class
Arm/Group | Bosentan | Pioglitazone
Number analyzed (Participants) | 1 | 1
NYHA class | 0 | 0

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | Bosentan | Pioglitazone
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1

LIMITATIONS AND CAVEATS:
Study terminated due to poor enrollment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No